CLINICAL TRIAL: NCT02371148
Title: Fase II Study With Bortezomib, Rituximab and Bendamustin-BRB- for Non-Hodgkin Lymphoplasmocytic Lymphoma/Waldenstrom Macroglobulinemia's Patients at First Relapse
Brief Title: Fase II Study With BRB for Non-Hodgkin Lymphoplasmacytic Lymphoma/Waldenstrom Macroglobulinemia's
Acronym: FIL_BRB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_BRB
Record Dates: First submitted 2015-02-13; First posted 2015-02-25 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Waldenstrom's Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib-Rituximab-Bendamustine (Experimental): Bortezomib-Rituximab-Bendamustine (BRB) combination in patients with relapsed/refractory lymphoplasmocytic/lymphoplasmocytoid lymphoma/Waldenstrom macroglobulinemia after one line of therapy.
  Interventions: Drug: Bortezomib-Rituximab-Bendamustine

INTERVENTIONS:
Drug: Bortezomib-Rituximab-Bendamustine — Bortezomib-Rituximab-Bendamustine Bortezomib: 1.3 mg/mq sc days 1, 8, 15, 22* Rituximab: 375 mg/sqm i.v. day 1** Bendamustine: 90 mg/sqm iv days 1-2 or days 2-3 according to institutional/physician choice Repeat cycles every 28 days for a total of 6 cycles *In case of toxicity is omitted
  **In cycles 1, in order to avoid tumor lysis syndrome, Rituximab will be given on day 8
  Other Names: BRB

SUMMARY:
This is a prospective, multicenter phase II trial designed to determine efficacy and safety of Bortezomib plus Rituximab plus Bendamustine in patients with relapsed/refractory Waldenstrom's Macroglobulinemia.

DETAILED DESCRIPTION:
The progression free survival (PFS) expected for lymphoplasmacytic/lymphoplasmocytoid lymphoma/Waldenstrom macroglobulinemia with the same characteristics indicated into the study and treated with standard Rituximab plus chemotherapy may be estimated to be 50% at 18 months.

The Investigators would consider a positive result to increase 18 months-PFS rate from 50 to 65%.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven diagnosis of Lymphoplasmacytic/cytoid lymphoma/Waldenstrom macroglobulinemia according to REAL/WHO Classification
* Relapsed/refractory disease after receiving one line chemotherapy (rituximab). If patients received bortezomib or bendamustine and have obtained a partial response lasting at least two years.
* Age >= 18
* Presence of at least one of the following criteria for the definition of active disease: Systemic symptoms or Hemoglobin less than 10 g/dL (due to lymphoma) or Platelets less than 100 x 109/L (due to lymphoma) or symptomatic splenomegaly or Bulky disease (>7 cm) or Hyperviscosity syndrome, peripheral neuropathy up to grade 1 (Waldenstrom's disease-related), hemolytic anemia, and immune complex vasculitis
* Life expectancy >6 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* left ventricular ejection fraction (LVEF) ≥45% or FS ≥37%
* Creatinine up to 1.5 x upper limit of normal
* Conjugated bilirubin up to 2 x upper limit of normal
* Alkaline phosphatase and transaminases up to 2 x upper limit of normal
* Written informed content

Exclusion Criteria:

* Patients who received bortezomib or bendamustine first-line therapy, that or haven't obtained at least partial response nor partial response lasting at least two years.
* Patients not agreeing to take adequate contraceptive precautions during and for at least 6 months after cessation of therapy
* History of other malignancies within 3 years prior to study entry except for: adequately treated carcinoma in situ of the cervix; basal or squamous cell skin cancer; low grade, early stage, localized prostate cancer treated surgically with curative intent; good prognosis ductal carcinoma in situ (DCIS) of the breast treated with lumpectomy alone with curative intent
* Medical condition requiring long term use (>1 months) of systemic corticosteroids
* Active bacterial, viral, or fungal infection requiring systemic therapy
* Peripheral neuropathy of any grade ≥ 2 [see Appendix Section A]
* Concurrent medical condition which might exclude administration of therapy
* Cardiac insufficiency (NYHA grade III/IV)
* Myocardial infarction within 6 months of entry on study
* Severe chronic obstructive pulmonary disease with hypoxemia
* Severe diabetes mellitus difficult to control with adequate insulin therapy
* Hypertension that is difficult to control
* Impaired renal function with creatinine clearance <30 ml/min
* HIV positivity HBV positivity with the exception of patients HbsAg and HBV-DNA negative and Ab anti-HB core positive (these patients need to receive prophylaxis with Lamivudine)
* HCV positivity with the exception of patients with HCV RNA negative
* Participation at the same time in another study in with investigational drugs are used
* Known hypersensitivity or anaphylactic reactions to murine antibodies or proteins
* Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent.
* Women in pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-06; Primary Completion 2017-11 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 18 months
  This is a prospective, multicenter phase II trial designed to determine efficacy and safety of Bortezomib plus Rituximab plus Bendamustine in patients with relapsed/refractory Waldenstrom's Macroglobulinemia. Primary Objective is to assess whether the experimental treatment achieves an absolute increase of PFS rate from 50 to 65% at 18 months with respect to the standard treatment. PFS is measured from the beginning of therapy to the date of disease progression, relapse or death from any cause.
  Patients without any relapse at the end of the follow-up will be censored at their last assessment date.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 2 years
  Overall response rate (ORR): a patient is defined as a responder if he has a complete or very good partial or partial response, evaluated in based on Waldenstrom macroglobulinemia consensus recommendations of the 6th International Workshop on Waldestrom's macroglobulinemia.
Overall Survival (OS) | 2 years
  Overall survival (OS): measured from the beginning of therapy to the date of death from any cause. Patients alive at the time of the final analysis will be censored at the date of the last contact. Minimum follow up time required for all patients will be 2 years.
Toxicity | 2 years
  Toxicity: severe, life- threatening, fatal (grade 3, 4 and 5)
Number of serious adverse events | 2 years
  Number of serious adverse events are defined according to "Common Terminology Criteria for Adverse Events" (CTCAE), version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Lorella Orsucci, MD, Principal Investigator — SC EMATOLOGIA - AO CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO; Giulia Benevolo, MD, Principal Investigator — SC EMATOLOGIA - AO CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO
Locations (23):
- Italy (23):
  - AO Riuniti Papardo Piemonte, Messina, ME
  - Centro di Riferimento Oncologico della Basilicata, Rionero in Vulture, PZ
  - AUSL di Ravenna, Ravenna, RA
  - A.O. Bianchi - Melacrino - Morelli, Reggio Calabria, RC
  - Nuovo Regina Margherita, Roma, RM
  - Uo Oncoematologia, Po "A.Tortora", Pagani, Salerno
  - Ospedale S. Giacomo di Castelfranco Veneto, Castelfranco Veneto, Treviso
  - A.O. SS. Antonio e Biagio e C. Arrigo, Alessandria
  - A.O. Universitaria Ospedali Riuniti - Ospedale Umberto I Di Ancona, Ancona
  - Centro di riferimento Oncologico - Oncologia Medica A, Aviano (PN)
  - A.O. Ospedale Degli Infermi, Biella
  - Ospedale Businco, Divisione di Ematologia, Cagliari
  - Area Vasta Romagna e IRST, Meldola (FC)
  - Irccs Ospedale Maggiore Policlinico Di Milano, Milan
  - A.O. Universitaria Policlinico Di Modena, Modena
  - Ospedale Maggiore Della Carita' - Scdu Ematologia, Novara
  - Ospedale San Martino, Asl Oristano- Ematologia, Oristano
  - Ematologia Policlinico San Matteo, Pavia
  - Ausl Di Piacenza, Piacenza
  - Ausl Di Rimini, Rimini
  - Ematologia 1 - A.O. Citta' Della Salute E Della Scienza Di Torino, Torino
  - Città della Salute e della Scienza SC Ematologia, Torino
  - Ematologia - OSPEDALE DI CIRCOLO E FONDAZIONE MACCHI, Varese

IPD SHARING:
Plan to Share IPD: Undecided